CLINICAL TRIAL: NCT07397897
Title: Intracranial EEG to Test How Noninvasive Stimulation Affects Hippocampal-dependent Memory
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB25-0756
Record Dates: First submitted 2026-01-20; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Memory Performance; Hippocampal Network Activity
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single pulse TMS stimulation (Experimental): The investigators will measure neural activity evoked by single pulses of Hippocampal Indirectly Targeted Stimulation (HITS). Stimulation intensity will vary to yield dose-response information. The investigators will also stimulate a control location. The investigators hypothesize that hippocampus/hippocampal-network intracranial EEG (iEEG) activity will respond to HITS, but not to control-location stimulation. Moreover, the selectivity of EPs will vary with HITS intensity, with very high intensities yielding less-selective (off-target) EP responses outside the hippocampal network. Findings consistent with these hypotheses would indicate that HITS directly impacts hippocampal and/or hippocampal-network neural activity
  Interventions: Other: Transcranial magnetic stimulation (TMS)
- Theta-burst TMS stimulation (Experimental): During task-free periods (fixation cross), HITS will be delivered in a theta-burst rhythm, versus two control non-theta rhythms and no-stimulation control. The investigators will test whether HITS entrains theta in the period immediately following 2-s trains of each condition. The investigators hypothesize that theta-burst HITS will entrain endogenous hippocampal and hippocampal-network theta more than control stimulation. Stimulation will also be delivered within a memory encoding task using naturalistic visual scenes. The investigators hypothesize that hippocampal theta entrainment by HITS will significantly increase during encoding relative to task-free periods, and that this effect will be selective versus the control stimulation conditions. Further, the investigators hypothesize that theta-burst HITS will improve memory relative to the control conditions. Such findings would indicate that HITS influences memory-related hippocampal theta activity.
  Interventions: Other: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Other: Transcranial magnetic stimulation (TMS) — Study conditions will involve different parameters for electrical stimulation delivered using non-invasive TMS.

SUMMARY:
Human intracranial electroencephalography (EEG) can provide brain-activity correlates of memory with high spatial and temporal resolution. This project will test functional relevance of these neural signals for memory behavioral performance using a novel noninvasive stimulation method. Findings will advance understanding of brain mechanisms for memory, as is needed to accelerate progress in the treatment of memory disorders.

DETAILED DESCRIPTION:
This exploratory project merges noninvasive brain stimulation with invasive/neurosurgical electrophysiological recordings in humans to identify mechanisms for how stimulation targeting the hippocampal network affects episodic memory performance. Hippocampal network dysfunction is associated with episodic memory impairments in a variety of neurologic and psychiatric disorders. Core regions of this network such as the hippocampus are too deep within the brain to be directly affected by well-validated noninvasive neuromodulation approaches. Hippocampal Indirectly Targeted Stimulation ("HITS") addresses this limitation by targeting the hippocampus indirectly via stimulation-accessible neocortical hippocampal-network locations, to which patterned transcranial magnetic stimulation is applied. HITS reliably improves episodic memory performance and increases fMRI activity of the hippocampal network, including the hippocampus. However, it is not clear how HITS affects neural activity to produce these effects. Memory performance is supported by spatiotemporally coordinated neural activity of the hippocampal network, such as in synchronization of thetafrequency band oscillatory activity. The investigators hypothesize that HITS directly influences this coordinated activity within the hippocampal network. Alternatively, HITS could have a variety of nonspecific, indirect, or neuromodulatory effects that are not necessarily specific to the hippocampal network. Intracranial EEG (iEEG) recorded from multi-contact depth macroelectrodes in patients undergoing neurosurgical procedures provides the required temporal and spatial precision needed to test the hypothesis that HITS directly impacts hippocampal network activity. The investigators therefore will perform HITS in patients undergoing iEEG. The investigators will determine the impact of HITS on activity of the hippocampal network versus on off-target brain areas. To test whether HITS influences the coordination of theta-band oscillatory activity that is especially important for memory, the investigators will use a stimulation rhythm that should maximally affect this activity (theta-burst patterned stimulation) versus control rhythms and will administer HITS during a memory task versus during task-free periods. This is an ideal exploratory project because HITS-iEEG has a strong scientific rationale but involves many technical and logistical challenges yet to be solved. Success could motivate highly impactful research using HITS-iEEG. For example, understanding neural mechanisms of how HITS improves episodic memory could illuminate how to achieve memory enhancement via other methods, such as by deep-brain stimulation, by portable noninvasive electrical stimulation methods, or by next-generation noninvasive stimulation technologies. This future research would have strong scientific potential, in providing stimulation-based causal tests of brain-behavior relationships for memory. Findings could motivate brain stimulation therapy for neurological and psychiatric memory disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years old
* Native English speakers
* Normal or corrected-to-normal near and far vision

Exclusion Criteria:

-iEEG electrode placement in area of parietal lobe that will interfere with placement of TMS coil for HITS stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Power of theta-band hippocampal electroencephalography (iEEG) activity | Measured while research activities are being completed, including during stimulation and the performance of the task . Measurement will take 2 to 4 hours on a single day.
  Power of theta-band hippocampal iEEG activity will be recorded and used to measure local brain electrical activity evoked by task conditions
Electroencephalography (iEEG) activity between hippocampus and the stimulated electrode | Measured while research activities are being completed, including during stimulation and the performance of the task . Measurement will take 2 to 4 hours on a single day.
  iEEG is used to measure local brain electrical activity evoked by task conditions. iEEG will be recorded and analyzed to determine the synchrony of iEEG activity between hippocampus and the stimulated electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Voss, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No